CLINICAL TRIAL: NCT06403332
Title: Study of the Drivers of Late Diagnosis of Alcohol Related Diseases, Alone or in Combination With Metabolic Dysfunconal Associated Fatty Liver Disease, Implementation and Evaluation of Itnerventions to Reduce Its Burden.
Acronym: StopALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Pompeu Fabra (Other); IDIAPJgol (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PR(AG)30/2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Alcohol-related Liver Disease; Alcohol Use Disorder; Metabolic and Alcohol Related/Associated Liver Disease; Metabolic Disfunction Associated Steatotic Liver Disease
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A intervention (Experimental)
  Interventions: Behavioral: brief intervention
- Cohort A non intervention (No Intervention)
- Cohort B intervention (Experimental)
  Interventions: Behavioral: brief intervention
- Cohort B no intervention (No Intervention)
- Control grup no significant liver disease (No Intervention)
- Control group MASLD (No Intervention)
- Control group decompensated ArLD (No Intervention)

INTERVENTIONS:
Behavioral: brief intervention — The intervention for cohort A (intervention arm) based on brief intervention on alcohol consumption performed by a psycologist, medical visit peformed by an hepatologist including assessment of underlying liver disease with non invasive test (i.e Fibroscan and lab work).
  Other Names: Diangostic test; Hepatology evaluation
  Arms: Cohort A intervention; Cohort B intervention

SUMMARY:
Excessive alcohol use is a leading risk factor for preventable disability and death. Alcohol-related liver disease (ALD) is one of the better-known detrimental consequences of alcohol abuse and is the main cause of disability-adjusted life years (DALYs) in European adults. ALD is the main cause of cirrhosis globally and is responsible for 60% of cirrhosis in Europe and North America.

Importantly, another etiology of liver disease is on the rise due to the epidemics of obesity and diabetes mellitus in Western countries, i.e., metabolic dysfunction associated fatty liver disease (MAFLD). ALD and MAFLD are largely shaped by social determinants of health (SDH) and lead to mounting health inequalities. Moreover, ALD is subject to strong stigmatization, particularly amongst women, which often leads to lack of inquiry by health professionals. Alone or in combination (MAFLD-OH), both diseases represent a challenge for epidemiologists, clinicians and policy makers in charge of health systems' organization. One of the hurdles to reduce the burden of ALD is the lack of early detection of asymptomatic liver disease among patients with alcohol use disorder (AUD) and heavy drinkers. The only measure that has been proven effective in any phase of the disease is to either stop, compensate, or reverse the liver disease progression, is alcohol abstinence. We hypothesize that establishing effective screening programs to identify patients with ALD and related disorders, coupled with effective treatment will lead to more positive outcomes in prognosis. The central aim of the StopALD Project is to identify patients with advanced ALD during the asymptomatic phases of the disease, as well as identifying the factors related with the lack of early detection to better implement interventions so to tackle both the lack of early detection of ALD and heavy drinking patterns among young people before ALD occurs.

ELIGIBILITY:
Never decompensated patients with ArLD suspicion

* Age over 30
* Diagnosis of AUD identified by the AUDIT test or excessive alcohol consumption, i.e., suspicion of current or recent (within one year) AUD or persistent alcohol intake of more than 40 g/daily for women and 60 g/daily for men based on medical history or self-reported history of excessive alcohol use, stigmata of alcohol use on physical exam, liver chemistry abnormalities, and/or alcohol-induced organ involvement other than decompensated liver disease
* Alanine (ALT) and aspartate aminotransferases (AST) <5 times upper normal limit
* Bilirubin <3 mg/dL or/and
* AST/ALT ratio >1.5 or/and
* GGT >100 mg/dL • Patients with a past history of decompensated advanced liver disease (i.e., episodes of jaundice, ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome) or known HCC
* Patients with severe extrahepatic disease or terminal illness

Young patients with risk alcohol intake and without liver disease

* Age between 18-30 years
* Diagnosis of AUD identified by the AUDIT test or for whom there is a high suspicion of current or recent (within one year) AUD or persistent alcohol intake of more than 40 g/daily for women and 60 g/daily for men based on medical history or self-reported history of excessive alcohol use, stigmata of alcohol use on physical exam and/or alcohol-induced organ involvement other than decompensated liver disease
* Normal liver test including AST, ALT, bilirubin and GGT. • Patients with a past history of decompensated advanced liver disease (i.e., episodes of jaundice, ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome) or known HCC
* Patients with severe extrahepatic disease or terminal illness

Previously or currently decompensated patients • Age over 30

* Diagnosed ALD with a current or previous liver-related decompensation (i.e., ascites or edemas, hepatic encephalopathy, hepatocellular carcinoma, upper gastrointestinal bleeding, spontaneous bacterial peritonitis or alcoholic hepatitis) • Terminal illness with less than 6 months live expectancy (except advanced hepatocellular carcinoma)
* Previous liver transplant recipient

Patients without significant liver disease

* Age over 30
* Alcohol intake of <10g per day without current or previous AUD or heavy alcohol intake • Significant liver pathology MASLD patients with a maximum alcohol intake of 20g per day.
* Age over 30
* Alcohol intake (<20g/day in women and <30g/day in men),
* Patients with obesity and/or diabetes mellitus type 2 and/or metabolic syndrome defined by the presence of two or more of the Eslam et al. criteria. • Patients with a past history of decompensated advanced liver disease (i.e., episodes of jaundice, ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome) or known HCC
* Patients with severe extrahepatic disease or terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-06-06 (Estimated); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
efficacy of medical interventional and psychologist | 1.5 years
  To assess the efficacy of medical intervention including a hepatology visit, brief intervention and counseling provided by a psychologist as well as the non-invasive assessment of underlying fibrosis degree (Fibroscan improvement of 2 or more points) on alcohol abstinence (assesses by autoreport number of standard units of alcohol) and relapses compared to current standard of care.
to assess the efficacy of an in-situ psychologist counseling including a motivational interview among young patients with heavy drinking on alcohol abstinence and relapses compared to current SOC | 1.5
  to assess the efficacy of an in-situ psychologist counseling including a motivational interview among young patients with heavy drinking on alcohol abstinence and relapses compared to current SOC (alcohol intake assessed by number of standard drinks)

SECONDARY OUTCOMES:
to assess the impact of the intervention on the underlying liver disease (fibrosis and steatosis degree and rate of complications/decompensations). | 1.5 years
  to assess the impact of the intervention on the underlying liver disease (fibrosis and steatosis degree and rate of complications/decompensations). Fibrosis assessed by Fibroscan fibrosis improvement defined as improvement of 2 or more points in the fibroscan. Liver events (i.e hepatic encephalopathy, ascites, edemas, upper gastrointestinal bleeding, alcohol associated hepatitis)
to investigate the prevalence of MAFLD-OH amongst these patients and whether metabolic risk factors increase the prevalence and severity at diagnosis of advanced liver fibrosis in patients with AUD or excessive alcohol intake | 1.5 years
  to investigate the prevalence of MAFLD-OH amongst these patients and whether metabolic risk factors increase the prevalence and severity at diagnosis of advanced liver fibrosis in patients with AUD or excessive alcohol intake. Severity of Fibrosis assessed by Fibroscan (severe disease Fibroscan > 8, % of severe disease between ALD group and MAFLD+OH)
to identify the risk factors associated to the late diagnosis of advanced liver disease in patients with compensated vs. decompensated ALD | 1.5 years
  to identify the risk factors associated to the late diagnosis of advanced liver disease in patients with compensated vs. decompensated ALD. (Specific design questionaries with socieconomical, mental health, educational factors)
to identify the risk factors associated to the late diagnosis of AUD in young population under 30yo | 1.5 years
  to identify the risk factors associated to the late diagnosis of AUD in young population under 30yo (Specific design questionaries with socieconomical, mental health, educational factors)
to analyze the associations between sociocultural determinants of alcohol-related issues in the healthcare system and the late diagnosis of AUD, excessive alcohol intake and ALD | 2 years
  to analyze the associations between sociocultural determinants of alcohol-related issues in the healthcare system and the late diagnosis of AUD, excessive alcohol intake and ALD (Specific design questionaries with socieconomical, mental health, educational factors)
to evaluate the cost-effectiveness and cost-equity of the proposed interventions to assess the late diagnosis of alcohol excessive intake and alcohol-related disease | 2 years
  to evaluate the cost-effectiveness and cost-equity of the proposed interventions to assess the late diagnosis of alcohol excessive intake and alcohol-related disease

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - University Hospital Vall d'Hebron, Barcelona